CLINICAL TRIAL: NCT06791330
Title: A Type 1 Diabetes Genetic Risk Score Discriminates Between Type 1 Diabetes and Type 2 Diabetes in Chinese
Brief Title: Genome-wide Association Study of Different Types of Diabetes and Construction of Genetic Risk Score
Status: Completed | Type: Observational
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Yang Xiao, Professor, Department of Metabolism and Endocrinology, Institute of Metabolism and Endocrinology, National Clinical Research Center for Metabolic Diseases, Second Xiangya Hospital, Central South University, Second Xiangya Hospital of Central South University
Other Study IDs: 2019GRS
Record Dates: First submitted 2025-01-20; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; genetic risk score; genome-wide association study; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Genetic Risk Score; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples were directly stored in a -80℃ freezer after sampling. DNA was extracted following the manufacturer's protocol. DNA was fragmented to construct a paired-end library by using a Covaris M220 sonicator. Samples were sequenced on the Illumina platform according to the standard protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Controls: Controls were defined as individuals without diabetes or a family history of diabetes within the same geographic area who had normal oral glucose tolerance test results
- Type 1 diabetes: All diagnoses for diabetes were required to adhere to the 1999 World Health Organization diabetes diagnosis criteria. Type 1 diabetes mellitus patients needed to meet specific criteria, including insulin dependence in the first 6 months and the presence of at least one designated islet autoantibody: glutamic acid decarboxylase antibody (GADA), protein tyrosine phosphatase antibody (IA-2A) and zinc transporter 8 antibody (ZnT8A).
- Type 2 diabetes: All diagnoses for diabetes were required to adhere to the 1999 World Health Organization diabetes diagnosis criteria. Type 2 diabetes mellitus patients also needed to show negative results for all three islet autoantibodies at onset, including glutamic acid decarboxylase antibody (GADA), protein tyrosine phosphatase antibody (IA-2A) and zinc transporter 8 antibody (ZnT8A).

SUMMARY:
To enhance the genetic profile of T1D patients in China and construct a Chinese-specific GRS and evaluated its ability to differentiate between T1D and controls, as well as between T1D and T2D.

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) is caused by autoimmune destruction of pancreatic beta cells, leading to severe insulin deficiency and requires life-long insulin therapy. Although traditionally viewed as a disease primarily affecting children and adolescents, recent epidemiological studies have demonstrated that over half of all new-onset T1D cases worldwide occur in adults. At present, methods to differentiate adult-onset T1D from T2D rely on the clinical phenotypes such as onset age and pattern, body mass index (BMI), C-peptide levels, and islet autoantibodies. However, the increasing rates of obesity in T1D, the presence of ketosis-prone T2D and idiopathic T1D, as well as unavailable autoantibody detection in some districts make it an increasing difficult challenge to accurately classify between adult-onset T1D and T2D. The discrimination of diabetes types is more challenging in the Chinese population due to the higher prevalence of early-onset T2D at a lower BMI than in European populations. Incorrectly identifying T1D as T2D can result in inadequate control of blood glucose levels, an elevated risk of ketoacidosis, and potentially severe and life-endangering complications. Therefore, it is crucial to search for new discriminative methods for different types of diabetes.

The genetic pathogenesis of T1D and T2D differ significantly, allowing for the differentiation of diabetes types based on genetic information. A T1D genetic risk score (GRS), comprising 31 HLA and non-HLA T1D-associated single nucleotide polymorphisms (SNPs), can be a useful tool to aid the discrimination between T1D and T2D. GRS2, which improved SNP capture of HLA DR-DQ risk including haplotype interactions and added non-DR-DQ loci, showed better discriminative power for the classification of diabetes type among multiethnic youth.

In this study, we employed GWAS to enhance the genetic profile of T1D patients in China. Additionally, our aim was to identify SNP tags for the HLA DR-DQ risk in the Chinese population, which could capture HLA DR-DQ risk and the interactions between these haplotypes. Using this information, we constructed a Chinese-specific GRS and evaluated its ability to differentiate between T1D and controls, as well as between T1D and T2D.

ELIGIBILITY:
Inclusion Criteria:

* All diagnoses for diabetes were required to adhere to the 1999 World Health Organization diabetes diagnosis criteria. Type 1 diabetes mellitus patients needed to meet specific criteria, including insulin dependence in the first 6 months and the presence of at least one designated islet autoantibody: glutamic acid decarboxylase antibody (GADA), protein tyrosine phosphatase antibody (IA-2A) and zinc transporter 8 antibody (ZnT8A). Type 2 diabetes mellitus patients also needed to show negative results for all three islet autoantibodies at onset. Controls were defined as individuals without diabetes or a family history of diabetes within the same geographic area who had normal oral glucose tolerance test results.

Exclusion Criteria:

* Subjects with the following conditions were excluded: severe gastrointestinal, cardiovascular, cerebrovascular, liver or kidney diseases; other autoimmune diseases; a history of gastrointestinal surgery; tumours; pregnancy; treatments with oral hypoglycaemic agents or immunomodulators; and use of probiotics, prebiotics or antibiotics within one month.

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects in these three groups were matched by age and sex.
Sampling Method: Probability Sample
Enrollment: 7000 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2024-04 (Actual); Study Completion 2024-04 (Actual)

PRIMARY OUTCOMES:
Identified single nucleotide polymorphisms that reach genome-wide significance | at baseline
  Single nucleotide polymorphisms should reach the genome-wide significance，which is defined as a P value of smaller than 5e-8.